CLINICAL TRIAL: NCT02008656
Title: A Phase II Multicenter Randomized Trial Evaluating 3-year Disease Free Survival in Patients With Locally Advanced Rectal Cancer Treated With Chemoradiation Plus Induction or Consolidation Chemotherapy and Total Mesorectal Excision or Non-operative Management
Brief Title: Trial Evaluating 3-year Disease Free Survival in Patients With Locally Advanced Rectal Cancer Treated With Chemoradiation Plus Induction or Consolidation Chemotherapy and Total Mesorectal Excision or Non-operative Management
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Colon and Rectal Surgery Inc. (Industry); The Cleveland Clinic (Other); John Muir Health (Other); Oregon Health and Science University (Other); St. Joseph Hospital of Orange (Other); University of California, Irvine (Other); University of California, San Francisco (Other); University of Chicago (Other); University of South Florida (Other); University of Vermont (Other); University of Washington (Other); Medstar Health Research Institute (Other); Washington University School of Medicine (Other); Creighton University Medical Center (Other); The Methodist Hospital Research Institute (Other); University of Rochester (Other); University of Virginia (Other); St. Paul's Hospital (Unknown); St. Joseph, Florida (Unknown); Cleveland Clinic Florida (Other); University of Colorado, Denver (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-213
Record Dates: First submitted 2013-11-27; First posted 2013-12-11 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: CAPECITABINE (ORAL); FLUOROURACIL; LEUCOVORIN; OXALIPLATIN; Total mesorectal excision; Chemoradiation therapy; Total neoadjuvant therapy; 13-213
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Capecitabine; Radiotherapy, Intensity-Modulated

ARMS (2):
- INCT (Experimental): Arm 1 will receive chemotherapy before chemoradiation. This is called induction neoadjuvant chemotherapy arm (INCT). The neoadjuvant chemotherapy regimen is prescribed specifically as 8 cycles of FOLFOX or 5 cycles of CapeOX over a period of approximately 15-16 weeks. Endoscopic exam (2-4 wks) after chemotherapy. If stable or response then pt will have radiation with either 5-FU or capecitabine.
  Interventions: Drug: Oxaliplatin (OXAL); Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin; Drug: Capecitabine (Xeloda®); Radiation: intensity modulated radiotherapy (IMRT); Behavioral: Quality of Life Questionnaires; Procedure: DRE-Endoscopy
- CNCT (Experimental): Arm 2 will receive chemoradiation before chemotherapy This is called the consolidation neoadjuvant chemotherapy arm (CNCT). Pt will have 6 weeks of chemoradiation therapy. Along with the radiation the pt will receive either 5-FU or capecitabine. 2-4 weeks after pt will have endoscopic exam and if stable or response pt will have will have 8 cycles of FOLFOX or 6 cycles of CapeOX.
  Interventions: Drug: Oxaliplatin (OXAL); Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin; Drug: Capecitabine (Xeloda®); Radiation: intensity modulated radiotherapy (IMRT); Behavioral: Quality of Life Questionnaires; Procedure: DRE-Endoscopy

INTERVENTIONS:
Drug: Oxaliplatin (OXAL)
Drug: 5-Fluorouracil (5-FU)
Drug: Leucovorin
Drug: Capecitabine (Xeloda®)
Radiation: intensity modulated radiotherapy (IMRT)
Behavioral: Quality of Life Questionnaires
Procedure: DRE-Endoscopy

SUMMARY:
The study is designed to test the hypothesis that patients with Locally advanced rectal cancer ( LARC) treated with Total neoadjuvant therapy (TNT) and Total mesorectal excision (TME) or Non-operative management (NOM) will have an improved 3-year disease-free survival (DFS) compared to patients with similar tumors treated with Chemoradiation therapy (CRT), Total mesorectal excision (TME) and Adjuvant chemotherapy (ACT).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the rectum
* Clinical Stage II (T3-4, N-) or Stage III (any T, N+) based on MRI
* Rectal tumor at baseline which would be considered to require complete TME
* No evidence of distant metastases
* No prior pelvic radiation therapy
* No prior chemotherapy or surgery for rectal cancer
* Age ≥ 18 years The minimum legal age of consent for select Canadian provinces is 19
* No active infections requiring systemic antibiotic treatment (oral antibiotics are acceptable at the discretion of the treating physician)
* ECOG Performance status 0-2
* Women with childbearing potential (WOCBP) who are negative for pregnancy test (urine or blood) and who agree to use effective contraceptive method. A woman of childbearing potential is defined of one who is biologically capable of becoming pregnant. Reliable contraception should be used from trial screening and must be continued throughout the study.
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study. Patients who do not read or understand English are eligible and may be consented according to institutional and federal regulations.
* ANC > 1.5 cells/mm3, HGB > 8.0 gm/dl, PLT > 150,000/mm3 total bilirubin ≤ 1.5 x ULN (except in patients with Gilbert's Syndrome who must have total bilirubin ≤ 3.0 x ULN), AST≤ 3 x ULN, ALT ≤ 3 x ULN.

Exclusion Criteria:

* Recurrent rectal cancer
* Primary unresectable rectal cancer. A tumor is considered unresectable when invading adjacent organs and an en block resection will not achieve negative margins.
* Creatinine level greater than 1.5 times the upper limit of normal.
* Patients who have received prior pelvic radiotherapy.
* Patients who are unable to undergo an MRI.
* Patients with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA, or CVA.
* Patients with a history of venous thrombotic episodes such as deep venous thrombosis, pulmonary embolus occurring more than 6 months prior to enrollment may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Similarly, patients who are anticoagulated for atrial fibrillation or other conditions may participate, provided they are on stable doses of anticoagulant therapy.
* Other Anticancer or Experimental Therapy. No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matrix metalloprotease inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibody or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
* WOCBP who are unwilling or unable to use an acceptable method of avoiding pregnancy for the entire study period.
* Women who are pregnant or breast-feeding.
* Patients with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study.
* Patients with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 years
  3-year DFS will be defined as the percentage of patients alive without recurrence of disease at 3 years measured from the date of randomization

SECONDARY OUTCOMES:
major adverse events | 3 years
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Garcia Aguilar, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (26):
- United States (26):
  - University of California, Irvine, Irvine, California
  - St. Joseph Hospital, Orange, California
  - University of California San Francisco, San Francisco, California
  - John Muir Health, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University Of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Northville, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - CHI Heath Bergan Mercy, Omaha, Nebraska
  - Colon and Rectal Surgery, Incorporated, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Derived] Manca P, Chen CT, Shah F, Lee C, Domenico D, Omer D, Gonzalez S, De Bruijn I, Ahuno S, Chatila WK, Darmofal M, Tavassoly I, Widman AJ, Berger MF, Loomis B, Papaemmanuil E, Yaeger R, Zviran A, Garcia-Aguilar J, Sanchez-Vega F. Ultrasensitive ctDNA monitoring for organ preservation in patients with locally advanced rectal cancer. NPJ Precis Oncol. 2025 Dec 11;10(1):8. doi: 10.1038/s41698-025-01208-w. PMID 41381715
- [Derived] Williams H, Omer DM, Thompson HM, Lin ST, Verheij FS, Miranda J, Yuval JB, Buckley J, Marco MR, Qin LX, Dombroski DA, Kedar R, Oto A, Korngold E, Veniero JC, Gandhi S, Krishnaraj A, Jagtiani M, Ohanian K, Vu D, Hope TA, Lee S, Wasnik AP, Madhuripan N, Gollub MJ, Garcia-Aguilar J; OPRA Consortium. MRI Predicts Residual Disease and Outcomes in Watch-and-Wait Patients with Rectal Cancer. Radiology. 2024 Sep;312(3):e232748. doi: 10.1148/radiol.232748. PMID 39225603
- [Derived] Thompson HM, Omer DM, Lin S, Kim JK, Yuval JB, Verheij FS, Qin LX, Gollub MJ, Wu AJ, Lee M, Patil S, Hezel AF, Marcet JE, Cataldo PA, Polite BN, Herzig DO, Liska D, Oommen S, Friel CM, Ternent CA, Coveler AL, Hunt SR, Garcia-Aguilar J; OPRA Consortium. Organ Preservation and Survival by Clinical Response Grade in Patients With Rectal Cancer Treated With Total Neoadjuvant Therapy: A Secondary Analysis of the OPRA Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2350903. doi: 10.1001/jamanetworkopen.2023.50903. PMID 38194231
- [Derived] Verheij FS, Omer DM, Williams H, Lin ST, Qin LX, Buckley JT, Thompson HM, Yuval JB, Kim JK, Dunne RF, Marcet J, Cataldo P, Polite B, Herzig DO, Liska D, Oommen S, Friel CM, Ternent C, Coveler AL, Hunt S, Gregory A, Varma MG, Bello BL, Carmichael JC, Krauss J, Gleisner A, Guillem JG, Temple L, Goodman KA, Segal NH, Cercek A, Yaeger R, Nash GM, Widmar M, Wei IH, Pappou EP, Weiser MR, Paty PB, Smith JJ, Wu AJ, Gollub MJ, Saltz LB, Garcia-Aguilar J. Long-Term Results of Organ Preservation in Patients With Rectal Adenocarcinoma Treated With Total Neoadjuvant Therapy: The Randomized Phase II OPRA Trial. J Clin Oncol. 2024 Feb 10;42(5):500-506. doi: 10.1200/JCO.23.01208. Epub 2023 Oct 26. PMID 37883738
- [Derived] Garcia-Aguilar J, Patil S, Gollub MJ, Kim JK, Yuval JB, Thompson HM, Verheij FS, Omer DM, Lee M, Dunne RF, Marcet J, Cataldo P, Polite B, Herzig DO, Liska D, Oommen S, Friel CM, Ternent C, Coveler AL, Hunt S, Gregory A, Varma MG, Bello BL, Carmichael JC, Krauss J, Gleisner A, Paty PB, Weiser MR, Nash GM, Pappou E, Guillem JG, Temple L, Wei IH, Widmar M, Lin S, Segal NH, Cercek A, Yaeger R, Smith JJ, Goodman KA, Wu AJ, Saltz LB. Organ Preservation in Patients With Rectal Adenocarcinoma Treated With Total Neoadjuvant Therapy. J Clin Oncol. 2022 Aug 10;40(23):2546-2556. doi: 10.1200/JCO.22.00032. Epub 2022 Apr 28. PMID 35483010
- [Derived] Shi DD, Mamon HJ. Playing With Dynamite? A Cautious Assessment of TNT. J Clin Oncol. 2021 Jan 10;39(2):103-106. doi: 10.1200/JCO.20.02199. Epub 2020 Oct 14. No abstract available. PMID 33052753
- [Derived] Smith JJ, Chow OS, Gollub MJ, Nash GM, Temple LK, Weiser MR, Guillem JG, Paty PB, Avila K, Garcia-Aguilar J; Rectal Cancer Consortium. Organ Preservation in Rectal Adenocarcinoma: a phase II randomized controlled trial evaluating 3-year disease-free survival in patients with locally advanced rectal cancer treated with chemoradiation plus induction or consolidation chemotherapy, and total mesorectal excision or nonoperative management. BMC Cancer. 2015 Oct 23;15:767. doi: 10.1186/s12885-015-1632-z. PMID 26497495
- [Derived] Garcia-Aguilar J, Chow OS, Smith DD, Marcet JE, Cataldo PA, Varma MG, Kumar AS, Oommen S, Coutsoftides T, Hunt SR, Stamos MJ, Ternent CA, Herzig DO, Fichera A, Polite BN, Dietz DW, Patil S, Avila K; Timing of Rectal Cancer Response to Chemoradiation Consortium. Effect of adding mFOLFOX6 after neoadjuvant chemoradiation in locally advanced rectal cancer: a multicentre, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):957-66. doi: 10.1016/S1470-2045(15)00004-2. Epub 2015 Jul 14. PMID 26187751
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/